CLINICAL TRIAL: NCT06106477
Title: Impact of Intermittent Fasting on Biomarkers of Inflammation and Health-Related Quality of Life: A Feasibility Trial for Women With HR+/HER2- Early Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sailaja Kamaraju, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00049422
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: intermittent fasting; obesity; overweight; breast cancer; hormone receptor positive; HER2-negative; human epidermal growth factor receptor 2-negative; HR-positive; HR+/HER2-; early breast cancer; adjuvant endocrine therapy
MeSH Terms: conditions — Breast Neoplasms; Intermittent Fasting; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intermittent Fasting (Experimental): Enrolled subjects are expected to start the study intervention after completion of definitive therapy and within three months of starting AET.
  Interventions: Behavioral: Intermittent Fasting

INTERVENTIONS:
Behavioral: Intermittent Fasting — Participants will be asked to adhere to a six-month intermittent fasting intervention, a daily-recurring dietary plan consisting of:
  * An approximately fourteen-hour nightly fasting period that is followed by
  * An approximately ten-hour eating period with their last meal of the day occurring between 17:00 (5:00 PM) and 21:00 (9:00 PM).

SUMMARY:
This single-arm study is designed to test the hypothesis that a six-month intermittent fasting (IF) intervention is feasible for patients to adhere to and improves health-related quality of life while subjects are on adjuvant endocrine therapy (AET).

DETAILED DESCRIPTION:
This is a single-arm pilot study (n=20) designed to evaluate whether a six-month intermittent fasting (IF) intervention, defined as a daily recurring fourteen-hour nightly fasting period, is feasible to adhere to and feasible to determine health outcomes in breast cancer patients with a body mass index (BMI) of ≥25 and who are scheduled to start adjuvant endocrine therapy (AET) after definitive therapy.

Subjects with hormone receptor positive, HER2-negative breast cancer will be enrolled into this study. Data on study feasibility, quality of life (QOL) and anthropometric measurements, and biomarkers will be collected and analyzed. After the study is completed, the investigators may also perform a post-hoc analysis on subjects who received adjuvant chemotherapy in combination with AET vs. AET alone.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients ≥ 18 years old who are willing to consent to an approximately 14-hour nighttime fasting period and an approximately 10-hour daytime eating period.
2. Histologically and/or cytologically confirmed diagnosis of estrogen receptor (ER) positive (ER+) and human epidermal growth factor receptor (HER) 2 negative (HER2-) localized breast cancer (stages I-III).

   1. Progesterone receptor positive or negative patients are allowed.
   2. Hormone receptor positivity is defined as ER positivity in at least 1% cells by immunohistochemistry (IHC). HER 2-negative breast cancer is defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization fluorescence in situ hybridisation (FISH), chromogenic in situ hybridization (CISH), or silver-enhanced in situ hybridization (SISH) test is required.
3. Body mass index (BMI) ≥ 25.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
5. Subject must be willing to start the intermittent fasting (IF) intervention within three months of starting adjuvant endocrine therapy (AET), or at the discretion of the treating providers, and within 30 days of study enrollment.
6. Subjects who received neoadjuvant or adjuvant chemotherapy must have recovered completely from chemotherapy-related side effects such as nausea/emesis as determined by the treating providers.
7. Subjects who received neoadjuvant endocrine therapy are eligible only after completion of their definitive surgery (i.e., when ready to start adjuvant endocrine therapy) and treating provider ensures complete closure and healing of surgical incisions.
8. Subjects who had adjuvant systemic chemotherapy within two to four weeks prior to starting the IF intervention are eligible if they have recovered from acute effects of prior therapy to near baseline as determined by the treating physician.
9. Subjects on a targeted therapy, such as cyclin-dependent kinase (CDK) 4/6 inhibitor, or selective estrogen receptor degrader (SERD), or other clinical trial participants in the adjuvant setting are eligible at the discretion of the treating physician.
10. Subject co-administered with any prescriptions that may cause dizziness, hypoglycemia, or hypotension need to be evaluated and deemed eligible by the treating physician.
11. Adequate hepatic, renal function and adequate bone marrow reserve as determined by the treating physician:

    1. aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × institutional upper limit.
    2. Total bilirubin ≤ 1.5 × upper limit of normal (ULN), except for subjects with Gilbert's syndrome who may be included if their total bilirubin is ≤ 3.0 × ULN and direct bilirubin ≤ 1.5 × ULN.
    3. alkaline phosphatase (ALP) ≤ 2.5 × institutional upper limit with exception that ALP of < 5 × ULN is acceptable in patients with elevated with ALP due to bone metastases (in the absence of liver metastases).
    4. Serum creatinine <1.5 × ULN.
    5. Absolute neutrophil count (ANC) ≥1000/µL.
    6. Subjects with lymphopenia are eligible at the discretion of the treating provider.

    i. Hemoglobin (Hb) ≥ 8g/dL. ii. Platelet count ≥ 100,000/µL.
12. Premenopausal woman:

    1. Premenopausal is defined as someone who has had menses at any time in the last 12 months. For premenopausal women who are eligible for this trial, the treating physician may choose to monitor ovarian function with laboratory tests e.g., follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol as clinically indicated to assess their menopausal status.
    2. Subjects must agree not to conceive throughout the study and must use accepted methods of contraception.
    3. Women of childbearing potential must have a negative pregnancy test within seven days of registration and or seven to 10 days prior to starting study treatment.
13. Subjects who have an atypical sleep-wake schedule or different eating schedules are eligible at the discretion of the study investigators and dietitians as long as they agree to nightly fasting.
14. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Subject who works late night shifts.
2. Subject that was or currently on a fasting diet (e.g., Keto diets), intervention, or an agent (e.g., Ozempic) for the explicit purpose of inducing weight loss in the past one year.
3. Subject with a history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa).
4. Presence of diabetes.
5. Presence of chronic dizziness or vertigo.
6. Presence of endocrine disorders prone to fluctuations in blood sugar (e.g., multiple neuroendocrine disorders, adrenal disorders, chronic hypoglycemia).
7. Poorly controlled neurological disorders as determined by the treating physician (e.g., epilepsy, Parkinson's disease, myasthenia gravis, syncope, pre-syncopal episodes).
8. Poorly controlled co-existing cardiac disease as determined by the treating physician, such as chronic hypotension, symptomatic congestive heart failure (New York Heart Association III-IV), unstable angina, arrythmia (e.g., atrial fibrillation, bradycardia, tachycardia).
9. History of heavy alcohol use as determined by the treating physician.
10. History of liver disease (cirrhosis, active hepatitis) or chronic renal disease.
11. Untreated or active infections such as hepatitis, human immunodeficiency virus (HIV), chronic unhealed infections.
12. Clinically significant illness or systemic disease as determined by the treating physician.
13. Recent hospitalization for a major illness, as determined by the treating physicians, within one month of enrollment.
14. Subject who is pregnant or breastfeeding. Subjects who become pregnant while on the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Subject adherence to the intermittent fasting schedule. | Six months
  This measure is the number of subjects who adhere to at least 80% of the intermittent fasting schedule (i.e., follow the schedule on average for at least eight out of 10 days) throughout the six-month intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Sailaja Kamaraju, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No